CLINICAL TRIAL: NCT01619956
Title: Osteotome Sinus Floor Elevation With or Without Grafting: a Randomized Controlled Study
Brief Title: Osteotome Sinus Floor Elevation With or Without Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); Shanghai Municipal Science and Technology Commission (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Junyu Shi, Chair of Oral and Maxillo-facial Implantology Department, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 663-2009
Record Dates: First submitted 2012-06-09; First posted 2012-06-15 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Dental Implants; Sinus Floor Augmentation; Bone Remodeling
Keywords: dental implants; osteotome sinus floor elevation; survival rate; sinus grafting; bone remodeling; RCT; radiographic analysis
MeSH Terms: interventions — Bone Transplantation; Bio-Oss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSFE with grafting (Experimental): OSFE with grafting (autogenous bone chips+xenograft material with a ratio of 1:4)
  Interventions: Device: SLA dental implants; Procedure: Osteotome sinus floor elevation; Procedure: Bone grafting
- OSFE without grafting (Active Comparator): OSFE without grafting. No grafting materials or autogenous bone chips were used.
  Interventions: Device: SLA dental implants; Procedure: Osteotome sinus floor elevation

INTERVENTIONS:
Device: SLA dental implants — Dental implant with surface modification.
  Other Names: Straumann, Straumann AG, Waldenburg, Switzerland
Procedure: Osteotome sinus floor elevation — After locating the implant position by a round bur, the pilot drilling was performed to the depth approximately 1-2 mm away from the sinus floor boundary according to the depth taken from the pre-surgical radiograph. The cortical part of the implant bed was further widened to either 3.5mm for 4.1mm implants or 4.2mm for 4.8mm implants. Then the elevation of the maxillary sinus was achieved and developed using osteotome (Straumann Osteotome Kit, Straumann AG, Waldenburg, Switzerland) by light malleting to create a "greenstick" fracture on the compact bone of sinus floor and to increase diameters gradually till the final depth. The sinus membrane was tested again for any perforation by Valsalva manoeuvre.
  Other Names: osteotome (Straumann Osteotome Kit, Straumann AG, Waldenburg, Switzerland)
Procedure: Bone grafting — the autogenous bone chips harvested during the drilling procedure was mixed up with Bio-Oss® in approximately 1: 4 ratio. And the mixture was placed into the 'socket' by osteotomes when elevating the sinus membrane until the final depth.
  Other Names: Bio-Oss®, Geistlich Pharma AG, Wolhusen, Switzerland.
  Arms: OSFE with grafting

SUMMARY:
The osteotome sinus floor elevation (OSFE) technique has been proved to be a predictable procedure for successful implant placement in posterior maxillae with limited bone height under sinus. OSFE is considered to be minimal invasive and minimal traumatic while having a limitation with regard to the residual bone height. According to the consensus conference in 1996, OSFE technique without bone grafting should be limited to RBH ranging from 7mm to 9mm. However, recent studies reported favorable results even with RBH of around 4mm. Moreover, there is still controversy regarding the necessity of a grafting material in order to maintain the space for new bone formation. Spontaneous bone formation was observed for OSFE without grafting by some researches.

Due to the lack of randomized controlled trial (RCTs), there is still no clear guideline for implant therapy in posterior maxillae with limited bone height. Neither is there any evidence to recommend or contraindicate the application of grafting materials in combination with OSFE.

The present RCT is aimed to evaluate the clinical success of OSFE with RBH of 2mm to 8 mm and to study whether the application of grafting material in combination with OSFE will be more favorable. The hypothesis is that the application of simultaneous grafting has no significant advantage in terms of clinical success. Spontaneous bone formation can be observed with implants placed using OSFE without grafting.

45 systemically healthy adults consecutively admitted for oral implant therapy will be randomly assigned to 2 test groups. Only one implant system will be used to minimize the implant-originated influencing factors. Bio-Oss® will be chosen as the bone substitute as it is currently the typical xenograft available. Autogenous bone will be also used as it is deemed as 'gold standard' for bone graft materials.

A panoramic radiograph and cone-beam CT should be taken to assess the pretreatment bone height under sinus. For T1 group, the autogenous bone chips harvested during the drilling procedure will be mixed up with Bio-Oss®. And the mixture is placed into the 'socket' by osteotomes when elevating the sinus membrane until the final depth. For T2 group, no grafting materials will be used. The subjects will be recalled for follow-up visits at 3 months, 6 months, 1 year, 2 years, 3 years,5years and 10 years after surgery for clinical and radiographic examination. Implant protrusion length, endo-sinus bone gain and crestal bone level will be measured on the radiographs using specialized software. ANOVA will be performed for the success rates of the 2 groups. Descriptive statistics will be used for the radiographic parameters.

The present study is aimed to provide preliminary evidence for an important clinical question that whether OSFE is predictable and reliable with RBH of less than 6mm and whether the application of grafting materials is necessary for this indication.

DETAILED DESCRIPTION:
1. Specific aims

   1. To evaluate the clinical success of implants placed in posterior maxillae with limited residual bone height (2mm to 8 mm) using OSFE with or without simultaneous grafting
   2. To study the influence of simultaneous grafting on the clinical success of dental implants in posterior maxillae using OSFE
   3. To observe the bone changes in the elevated space under sinus with or without grafting.

   The null hypothesis is that the application of simultaneous grafting has no significant advantage in terms of clinical success. Spontaneous bone formation can be observed with implants placed using OSFE without grafting.
2. Background and significance

Posterior maxillae commonly pose a challenge for successful dental implants due to the poor bone quality and insufficient bone quantity. Efforts have been made to allow successful implant placement in the posterior maxilla subject to limited bone height under the sinus. Approaches available now include the application of tilting implants, short implants, sinus floor elevation technique, etc. The osteotome sinus floor elevation (OSFE) technique, first introduced by Tatum in 1986, has been proved to be a predictable procedure. For OSFE, access to the sinus membrane is achieved through a crestal approach. Therefore, compared with window technique, OSFE is considered to be less invasive and less traumatic while having a limitation with regard to the residual bone height. According to the consensus conference in 1996, OSFE technique should be limited to RBH ranging from 7mm to 9mm. However, with the improvement of implant design and surgical technique, the high predictability of implant therapy has encouraged re-evaluation of this limitation. Favorable results have been reported with more compromised sites even with RBH of around 4mm. Moreover, there is controversy regarding the necessity of a grafting material in order to maintain the space for new bone formation. In a previous pilot study, 42 implants was placed in posterior maxillae with OSFE without bone grafting materials. The RBH ranged from 4mm to 8mm (average 6.36mm). The 5-month result also demonstrated predictable results.

But to date, there is still insufficient data regarding the clinical results of the implants in posterior maxilla with OSFE technique without grafting and it still remains to be elucidated the necessity of grafting with OSFE. And the lack of well-designed RCTs makes the level of evidence relatively low. In this context, therefore, the applicants attempt to assess the clinical success of dental implants placed in posterior maxillae using OSFE with or without grafting and to observe the endo-sinus bone changes specially for RBH of only 2mm to 8 mm.

C. Methods

Randomization Subjects will be allocated to the two groups using the random numbers table. Allocation will be equalized every 20 cases. One research assistant will perform the randomization.

Study visits and procedures Pretreatment Assessment (Baseline) History-taking and consent taking: A detailed examination should be taken to make sure that the subject should fulfill the inclusion criteria. The subject will read through and sign the consent form.

Examination: A detailed dental examination should be performed to assess the intended implant site, which should include the dimension of the edentulous site, the status of mucosa and the status of adjacent teeth.

Baseline: A panoramic radiograph and an cone-beam CT should be taken to assess the pretreatment bone height under sinus.

Surgical procedure (Surgical Day):

Local infiltration anesthesia is used for all the subjects. A midcrestal incision, with mesial and distal releasing incisions extending well up into the buccal fold is performed and a full-thickness muco-periosteal flap is reflected. A round bur (Φ2.3 mm) is first used to mark the implant positions. Then, a minimal pilot drilling (Φ2.2mm) is performed to the depth approximately1 mm away from the sinus floor boundary according to the depth taken from the panoramic radiograph or CT scan. The cortical part of the implant bed is further widened to either Φ3.5mm forΦ4.1mm implants or Φ 4.2mm for Φ4.8mm implants. At this stage, the integrity of the sinus membrane is examined using the Valsava manoeuvre. Then the elevation of the maxillary sinus is achieved using Φ2.8mm osteotome by light malleting to achieve the initial sinus upfracture and is developed with osteotomes of increasing diameters gradually till the final depth.

For group1 , the autogenous bone chips harvested during the drilling procedure was mixed up with Bio- Oss®. And the mixture is placed into the 'socket' by osteotomes when elevating the sinus membrane until the final depth.

No grafting materials will be used for group2. No profile drill is used for any of the cases. The implants are placed in the prepared osteotomy site using a hand ratchet without tapping. All implants are placed in sites using a nonsubmerged technique and in a one stage procedure.

Postoperative treatment Amoxicillin (Xinya Co., Shanghai, China, 500mg, 4 times a day for 7 days) and metronidazole (Xinyiwanxiang, Shanghai, China, 400mg, 3 times a day for 7 days) will be used. Nonsteroidal anti-inflammatory agents are prescribed for post-surgical analgesia. 0.12% chlorhexidine oral rinse was prescribed for 60 seconds 5-6 times a day for 14 days. Sutures were removed after 1 week.

Patients were not allowed to use any removable prostheses during healing period. Patients should avoid blowing the nose during the healing period.

Prosthetic Procedure (Prosthetic Day) The implants are allowed to heal for 6 months. Porcelain-fused-to-gold prostheses are attached to the implants 7 to 10 days after impression taking.

Follow-ups The subjects will be recalled for follow-up visits at 3 months, 6 months, 1 year, 2 years, 3 years, 5years and 10 years after surgery for clinical and radiographic examination.

Parameters examined

Radiographic parameters:

1. Baseline: Pretreatment bone height under sinus at the implant site (mesial and distal)
2. Surgical Day: Implant protrusion length (mesial and distal)
3. Prosthetic Day and Follow-ups: Endo-sinus bone gain (mesial and distal)
4. Prosthetic Day and Follow-ups: Crestal bone level (mesial and distal)

Clinical parameters:

1. Surgical day: Schneiderian membrane integrity
2. Follow-ups: Post-operative complications (e.g. nose bleeding, infection)
3. Follow-ups: Implant mobility
4. Follow-ups: Probing depth Data collection Radiographic data: A panoramic and intra-oral radiograph will be taken at follow-up visits. For intra-oral radiograph, parallel technique will be applied. One experienced staff at the department of radiology will be responsible for taking these radiographs. The parameters will be measured using the specialized software.

Clinical data: Dr. Huan-Huan Jiang and Dr. Shi-Chong Qiao, who are blind to which group the subjects belong to, will be responsible for clinical data collection.

Statistical analysis ANOVA will be performed for the success rates of the 3 groups. The criterion for significance was set at α=0.05 and β=0.20. The ANOVA is non-directional. Descriptive statistics will be used for the radiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* partial edentulism in the maxillary posterior region for at least 6 months from tooth loss
* residual bone height ranged from 2mm to 8mm (measured on pre-surgical radiograph)
* sufficient bone width in edentulous region
* systemic and local condition compatible with implant placement and sinus floor elevation
* willing to provide informed consent and capable to comply the study protocol.

Exclusion Criteria:

* uncontrolled diabetes mellitus or other systemic disorders
* uncontrolled periodontal conditions, endodontic lesions or other oral disorders
* heavy smokers (≥ 10 cigarettes per day)
* rhinitis or sinusitis
* insufficient residual bone quality to achieve implant stability
* previous implant installation or bone grafting at the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Endo-sinus bone gain at 6-month | 6-month follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of both groups were assessed on radiography.
Endo-sinus bone gain at 12-month | 12-month follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of both groups were assessed on radiography.
Endo-sinus bone gain at 24-month | 24-month follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of both groups were assessed on radiography.
Endo-sinus bone gain at 36-month | 36-month follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of both groups were assessed on radiography.
Endo-sinus bone gain at 60-month | 60-month follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of bothgroups were assessed on radiography.
Endo-sinus bone gain at 10-year | 10-year follow-up
  Radiographic assessment was conducted on periapical radiographs at every follow-up visit using paralleling technique. The endo-sinus bone gain of bothgroups were assessed on radiography.

SECONDARY OUTCOMES:
Surgical and post-surgical complications and discomfort | 3 hours after surgery
  The sinus membrane perforation was evaluated by the Valsalva manoeuvre during surgery. Other surgical and post-surgical complications including infection, haemorrhage, nasal bleeding, benign paroxysmal positional vertigo (BPPV), blocked nose were also recorded.
  The pain and discomfort reported by the patients were evaluated by visual analogue scales (VAS) in which 0 indicated "no pain or no discomfort" and 100 indicated "intolerable pain or maximum discomfort"

CONTACTS AND LOCATIONS:
Overall Officials: Hongchang Lai, Principal Investigator — Department of Oral and Maxillo-facial Implantology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Department of Oral and Maxillo-facial Implantology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Tan WC, Lang NP, Zwahlen M, Pjetursson BE. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. Part II: transalveolar technique. J Clin Periodontol. 2008 Sep;35(8 Suppl):241-54. doi: 10.1111/j.1600-051X.2008.01273.x. PMID 18724853
- [Background] Lai HC, Zhuang LF, Lv XF, Zhang ZY, Zhang YX, Zhang ZY. Osteotome sinus floor elevation with or without grafting: a preliminary clinical trial. Clin Oral Implants Res. 2010 May;21(5):520-6. doi: 10.1111/j.1600-0501.2009.01889.x. Epub 2010 Mar 11. PMID 20337666
- [Background] Lai HC, Zhang ZY, Wang F, Zhuang LF, Liu X. Resonance frequency analysis of stability on ITI implants with osteotome sinus floor elevation technique without grafting: a 5-month prospective study. Clin Oral Implants Res. 2008 May;19(5):469-75. doi: 10.1111/j.1600-0501.2007.01501.x. Epub 2008 Mar 26. PMID 18371099
- [Background] Pjetursson BE, Ignjatovic D, Matuliene G, Bragger U, Schmidlin K, Lang NP. Transalveolar maxillary sinus floor elevation using osteotomes with or without grafting material. Part II: Radiographic tissue remodeling. Clin Oral Implants Res. 2009 Jul;20(7):677-83. doi: 10.1111/j.1600-0501.2009.01721.x. PMID 19515059
- [Background] Bragger U, Gerber C, Joss A, Haenni S, Meier A, Hashorva E, Lang NP. Patterns of tissue remodeling after placement of ITI dental implants using an osteotome technique: a longitudinal radiographic case cohort study. Clin Oral Implants Res. 2004 Apr;15(2):158-66. doi: 10.1111/j.1600-0501.2004.00988.x. PMID 15008927
- [Background] Tetsch J, Tetsch P, Lysek DA. Long-term results after lateral and osteotome technique sinus floor elevation: a retrospective analysis of 2190 implants over a time period of 15 years. Clin Oral Implants Res. 2010 May;21(5):497-503. doi: 10.1111/j.1600-0501.2008.01661.x. PMID 20443802
- [Background] Nedir R, Nurdin N, Vazquez L, Szmukler-Moncler S, Bischof M, Bernard JP. Osteotome sinus floor elevation technique without grafting: a 5-year prospective study. J Clin Periodontol. 2010 Nov;37(11):1023-8. doi: 10.1111/j.1600-051X.2010.01610.x. Epub 2010 Aug 24. PMID 20735796
- [Derived] Qian SJ, Mo JJ, Si MS, Qiao SC, Shi JY, Lai HC. Long-term outcomes of osteotome sinus floor elevation with or without bone grafting: The 10-year results of a randomized controlled trial. J Clin Periodontol. 2020 Aug;47(8):1016-1025. doi: 10.1111/jcpe.13260. Epub 2020 May 6. PMID 31976567
- [Derived] Si MS, Zhuang LF, Gu YX, Mo JJ, Qiao SC, Lai HC. Osteotome sinus floor elevation with or without grafting: a 3-year randomized controlled clinical trial. J Clin Periodontol. 2013 Apr;40(4):396-403. doi: 10.1111/jcpe.12066. Epub 2013 Feb 21. PMID 23425152